CLINICAL TRIAL: NCT01999881
Title: Impacts of Exercise on Prognostic Biomarkers in Lung Cancer Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: UW13034; NCI-2013-02185 (Registry Identifier: NCI Trial ID); 2013-0752 (Other: Institutional Review Board); UW13034 (Other: University of Wisconsin Carbone Cancer Center); P30CA014520 (NIH); A534260 (Other: UW Madison); SMPH\MEDICINE\HEM-ONC (Other: UW Madison)
Record Dates: First submitted 2013-11-25; First posted 2013-12-03 (Estimated); Last update posted 2019-11-18 (Actual); Status verified 2016-02

CONDITIONS: Extensive Stage Small Cell Lung Cancer; Healthy, no Evidence of Disease; Limited Stage Small Cell Lung Cancer; Recurrent Non-small Cell Lung Cancer; Recurrent Small Cell Lung Cancer; Stage IA Non-small Cell Lung Cancer; Stage IB Non-small Cell Lung Cancer; Stage IIA Non-small Cell Lung Cancer; Stage IIB Non-small Cell Lung Cancer; Stage IIIA Non-small Cell Lung Cancer; Stage IIIB Non-small Cell Lung Cancer; Stage IV Non-small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Small Cell Lung Carcinoma

ARMS (2):
- Arm A (aerobic and exercise training) (Experimental): Patients and their support persons undergo a supervised combined aerobic exercise comprising walking, cycling, or video-based aerobics and strength training using resistance bands for 40 minutes 2 days a week at the UWHC and 3 days a week at home over 8 weeks.
  Interventions: Behavioral: exercise intervention; Procedure: quality-of-life assessment; Other: laboratory biomarker analysis
- Arm II (usual care) (Active Comparator): Patients and their support persons undergo the usual care over 8 weeks.
  Interventions: Procedure: standard follow-up care; Procedure: quality-of-life assessment; Other: laboratory biomarker analysis

INTERVENTIONS:
Behavioral: exercise intervention — Receive aerobic and exercise intervention
  Arms: Arm A (aerobic and exercise training)
Procedure: standard follow-up care — Receive usual care
  Arms: Arm II (usual care)
Procedure: quality-of-life assessment — Ancillary studies
  Other Names: quality of life assessment
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
This randomized pilot clinical trial studies exercise intervention in improving quality of life and exercise capacity and reducing inflammation and oxidative stress in patients with lung cancer and their support persons. Exercise therapy may help improve quality of life, may increase exercise capacity, and may reduce inflammation and oxidative stress in patients with lung cancer and their supporters.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine the effect of an eight-week exercise intervention on biomarkers of inflammation, oxidative stress, exercise capacity, and quality of life in lung cancer patients.

SECONDARY OBJECTIVES:

I. Determine the effect of an eight-week exercise intervention on markers of stress and quality of life in the support person of lung cancer patients.

OUTLINE: Participants are randomized to 1 of 2 arms.

ARM A: Patients and their support persons undergo a supervised combined aerobic exercise comprising walking, cycling, or video-based aerobics and strength training using resistance bands for 40 minutes 2 days a week at the University of Wisconsin Hospital and Clinic (UWHC) and 3 days a week at home over 8 weeks.

ARM B: Patients and their support persons undergo the usual care over 8 weeks.

ELIGIBILITY:
Inclusion Criteria:

* LUNG CANCER PATIENTS: A confirmed diagnosis of any stage lung cancer (non-small cell lung cancer [NSCLC] or small cell lung cancer [SCLC])
* LUNG CANCER PATIENTS: Can be receiving any type of treatment (chemotherapy, radiation therapy, both or neither) are eligible
* LUNG CANCER PATIENTS: Able to understand and read in English sufficiently to adequately complete informed consent to participate and to complete the questionnaires
* LUNG CANCER PATIENTS: For patients treated with curative intent, and who have not relapsed, they must be within 1 year of their diagnosis of lung cancer (determined by date of diagnostic pathology sample)
* SUPPORT PERSONS: Able to understand and read in English sufficiently to adequately complete informed consent to participate and to complete the questionnaires

Exclusion Criteria:

* LUNG CANCER PATIENTS: Symptomatic heart disease including congestive heart failure or arrhythmia
* LUNG CANCER PATIENTS: Documented myocardial infarction in the last three months
* LUNG CANCER PATIENTS: Central nervous system (CNS) metastases that results in impaired ability to participate in an exercise program at the discretion of the study physician
* LUNG CANCER PATIENTS: Any psychological or physical disease that would impair or prevent participation in an exercise program at the discretion of the study physician
* LUNG CANCER PATIENTS: Cognitive or reading impairments that would preclude them from completing questionnaires
* LUNG CANCER PATIENTS: Current participation in an exercise program
* SUPPORT PERSONS: Symptomatic heart disease including congestive heart failure or arrhythmia
* SUPPORT PERSONS: Documented myocardial infarction in the last three months
* SUPPORT PERSONS: Cognitive or reading impairments that would preclude them from completing questionnaires

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2013-12; Primary Completion 2015-07 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Change in biomarkers of inflammation | Baseline up to 8 weeks
  Descriptive statistics will be calculated and compared between the two treatment groups at baseline using unpaired t-tests and Chi-Square analyses. A two-way analysis of variance will be used to examine the effects of the treatment over time.
Change in oxidative damage as indicated by serum 8-hydroxydeoxyguanosine (8-oh-dG) | Baseline up to 8 weeks
  Descriptive statistics will be calculated and compared between the two treatment groups at baseline using unpaired t-tests and Chi-Square analyses. A two-way analysis of variance will be used to examine the effects of the treatment over time.
Change in time to walk 400 m | Baseline up to 8 weeks
  Descriptive statistics will be calculated and compared between the two treatment groups at baseline using unpaired t-tests and Chi-Square analyses. A two-way analysis of variance will be used to examine the effects of the treatment over time.
Change in physical well-being scores on the Functional Assessment of Cancer Therapy-Lung (FACT-L) | Baseline up to 8 weeks
  Descriptive statistics will be calculated and compared between the two treatment groups at baseline using unpaired t-tests and Chi-Square analyses. A two-way analysis of variance will be used to examine the effects of the treatment over time.
Change in functional well-being scores on the FACT-L | Baseline up to 8 weeks
  Descriptive statistics will be calculated and compared between the two treatment groups at baseline using unpaired t-tests and Chi-Square analyses. A two-way analysis of variance will be used to examine the effects of the treatment over time.

SECONDARY OUTCOMES:
Change in stress scores on the SF-36 | Baseline up to 8 weeks
  Descriptive statistics will be calculated and compared between the two treatment groups at baseline using unpaired t-tests and Chi-Square analyses. A two-way analysis of variance will be used to examine the effects of the treatment over time.
Change in quality-of-life scores on the SF-36 | Baseline up to 8 weeks
  Descriptive statistics will be calculated and compared between the two treatment groups at baseline using unpaired t-tests and Chi-Square analyses. A two-way analysis of variance will be used to examine the effects of the treatment over time.

CONTACTS AND LOCATIONS:
Overall Officials: Toby Campbell, Principal Investigator — University of Wisconsin, Madison
Locations (2):
- United States (2):
  - UW Health Oncology - 1 South Park, Madison, Wisconsin
  - University of Wisconsin, Madison, Madison, Wisconsin

REFERENCES:
- See also: University of Wisconsin Carbone Cancer Center — https://cancer.wisc.edu/